CLINICAL TRIAL: NCT04273048
Title: A Dietary and Exercise Intervention in Overweight and Obese Women Undergoing Fertility Treatment
Brief Title: The MOM TO BE Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Terminated due to slow accrual or other non-safety related issues.
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 260113
Record Dates: First submitted 2019-11-13; First posted 2020-02-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: This research will last up to 12 weeks. The participant will attend two research study visits and will be asked to donate oocytes and follicular fluid to the study team during their oocyte retrieval procedures. They will be randomized (like flipping a coin) to either a standard of care group or an intervention group. If they are in the intervention group, they will also be asked to follow a Mediterranean diet (all meals will be shipped to their home weekly) and exercise at least 3 times a week at a gym or at their house. If they are in the control group, they will follow the normal fertility clinic procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet and Exercise (Active Comparator): Group 1 = Diet Intervention group: They will be asked to follow a personalized diet during study period and record what they eat. The meal plan for this study is Mediterranean style and nutritionally complete for 8 to 12 weeks or until oocyte retrieval procedure. Exercise Intervention: Exercise 3 times/week at a gym of their choice or at home for 8 to 12 weeks or until oocyte retrieval procedure. Exercises will be light intensity and short duration at first and will gradually increase to moderate intensity and longer duration during the first 3 weeks. They will also be encouraged to walk an average 10,000 steps per day and wear a pedometer to monitor progress.
  Interventions: Other: Diet Intervention - Group 1; Other: Exercise Intervention - Group 1
- Standard Care (No Intervention): Group 2 = Standard: They will receive standard care from the Little Rock Fertility Center.

INTERVENTIONS:
Other: Diet Intervention - Group 1 — They will be provided with a Mediterranean diet plan.
  Arms: Diet and Exercise
Other: Exercise Intervention - Group 1 — They will be provided with an exercise plan to follow.
  Arms: Diet and Exercise

SUMMARY:
This research study is about the effects of diet and exercise in women undergoing fertility treatment.

DETAILED DESCRIPTION:
This study will randomize women who are undergoing fertility treatment and put them either in an intervention group or standard care. This study should help us learn if diet and exercise changes oocytes gene expression and follicular fluid content.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 - 45 kg/m2
* ≥ 21 years of age

Exclusion Criteria:

* Pre-existing conditions (e.g. sexual transmitted diseases) that will affect the outcomes of the study as determined by the principal investigator
* Current use of recreational drugs, tobacco, or alcohol
* Food allergies, intolerances or preferences which would interfere with compliance to the meal plan
* Contraindications to exercise
* Already meeting the physical activity guidelines (150 min moderate activity/week or 75 minutes of vigorous activity/week with resistance exercise on 2 or more days/week).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Oocyte gene expression profile | 8-12 weeks
  Oocyte gene expression
Follicular fluid content | 8-12 weeks
  Follicular fluid content

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fawcett K, Martinez A, Crimmins M, Sims C, Borsheim E, Andres A. Effect of a dietary and exercise intervention in women with overweight and obesity undergoing fertility treatments: protocol for a randomized controlled trial. BMC Nutr. 2021 Aug 17;7(1):51. doi: 10.1186/s40795-021-00454-y. PMID 34399856